CLINICAL TRIAL: NCT05621603
Title: Adapting and Testing an Intervention to Integrate Workforce Mental Health Into Pre-K-8 School Emergency Preparedness Via Shared Leadership and Peer Support
Brief Title: Workforce Mental Health Emergency Preparedness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado School of Public Health (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Courtney Welton-Mitchell, Clinical Assistant Professor, Colorado School of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-4190
Record Dates: First submitted 2022-11-04; First posted 2022-11-18 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Mental Health; Burnout, Psychological
MeSH Terms: conditions — Psychological Well-Being; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: We will employ a matched waitlist control comparison design. Schools (6) will be randomly assigned to either the training arm or the control arm. Schools assigned to the control arm will eventually receive the training.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training (Experimental): Participants receive the intervention, which is a training program.
  Interventions: Behavioral: Training
- Control (No Intervention): Participants do NOT receive the intervention, which is a training program. This is a waitlist control comparison model.

INTERVENTIONS:
Behavioral: Training — The proposed intervention for the school workforce draws on a mental health integrated disaster preparedness model, emphasizing peer support, developed and used successfully by our team working with communities experiencing multiple disasters.
  The 3 hour training is comprised of 4 modules - Module 1: Emergency Preparedness Module 2: Psychological Preparedness Module 3: Peer Support Module 4: Shared Leadership and Feedback Session
  Arms: Training

SUMMARY:
School leaders, staff, and teachers are tasked with keeping children safe from acts of violence, natural hazards and other emergencies while encouraging learning. Disaster plans are often developed without teacher involvement, resulting in limited knowledge of emergency preparedness, undermining buy-in and limited motivation to comply with safety protocols, including disaster drills. The lack of initial consultation and limited decision-making authority can also be sources of stress for teachers. Teachers and staff may experience anxiety about their roles and responsibilities in a crisis. This research project proposes that the key to enhancing emergency preparedness in this population is to incorporate 'psychological preparedness' within a disaster management framework. In other words, to provide the school workforce with awareness of their likely psychological response to threat and coping skills/strategies for management of that response. Importantly, workforce-focused mental health integrated approaches to emergency preparedness are likely to work best if implemented via peer support and shared leadership frameworks. This project involves adaptation and implementation of an integrated workforce mental health intervention into Pre-K-12 school emergency preparedness via shared leadership and peer support. This includes co-creating training curriculum with Pre-K-12 schools, labor organizations, and district officials, implementing and evaluating the impact of the intervention. A matched waitlist control comparison research design will be used with six Pre-K-12 schools. The hypothesized outcomes of the intervention are increases in H1: emergency preparedness climate; emergency preparedness specific H2: shared leadership; H3: peer support and social cohesion; H4: confidence (in emergency preparedness); and H5: psychological preparedness. The project also anticipates H6: increases in overall mental health and well-being, and H7: a reduction in emergency preparedness-specific burnout.

DETAILED DESCRIPTION:
The burden of poor physical and mental health is high in the Pre-K-8 school workforce. While school employees had lower than average non-fatal occupational injury and illness rates overall in 2019, they had significantly higher rates of injury due to violence (35.5 per 10,000 FTEs vs overall 4.4 per 10,000 FTEs; R100).In addition, mental health needs are higher among teachers than the general population and are a contributing factor to burnout and teacher/staff turnover. Recent estimates of the burden of the COVID-19 pandemic has shed light on the impact that an emergency can have on the education sector workforce, with teachers feeling ill-equipped to adapt to increased expectations associated with safety protocols, online learning and student mental health. Thus, there is an urgent need to enhance emergency preparedness amongst the schools' workforce and a specific need to ensure that they can respond to the needs of others while maintaining their own mental health.

Nearly all public schools have emergency preparedness plans in place. However, disaster plans are often developed at the district level without teacher and staff involvement. This can result in limited knowledge of emergency preparedness and can undermine buy-in and decrease motivation to comply with safety protocols, including disaster drills. Furthermore, the lack of initial consultation and limited decision making authority can be a source of stress among teachers. Teachers and staff may experience anxiety about their roles and responsibilities in a crisis, including keeping themselves and children safe and managing expectations from parents and other stakeholders. It is reasonable to expect some teachers and staff to have strong reactions to drills for active shooter events, weather emergencies and/or disease outbreaks. Staff with a history of trauma exposure, at the school of elsewhere, may be especially vulnerable. Investigators propose that the key to enhancing emergency preparedness in this population is to incorporate 'psychological preparedness' within a disaster management framework. In other words, to provide the school workforce with awareness of their likely psychological response to threat and coping skills/strategies for management of that response. Importantly, such workforce-focused mental health integrated approaches to emergency preparedness are likely to work best if implemented via peer support and shared leadership frameworks. Such approaches have the potential to enhance the effectiveness and sustainability of existing efforts.

Investigators hypothesize that a half-day training intervention for Pre-K-12 schools that emphasizes integration of psychological preparedness with emergency preparedness, via shared leadership and peer support, will increase - H1: the emergency preparedness climate; H2: shared leadership for emergency preparedness; H3: peer support and social cohesion associated with emergency preparedness; H4: confidence (in emergency preparedness); and H5: psychological preparedness. Investigators also hypothesize that investigators will observe (H6) an increase in overall mental health and wellbeing, and a reduction in (H7) emergency preparedness-specific burnout. Thus, the impact of this intervention will be on the school workforce's capability to respond to emergencies while maintaining their well-being.

Specific Aim 1: Adapt and implement an integrated workforce mental health intervention into Pre-K-8 school emergency preparedness via shared leadership and peer support.

* Review emergency preparedness plans/drills and mental health supports at 6 Pre-K-12 schools
* Co-create training curriculum with participating schools and district officials (N = 64, 6 focus groups with 36 participants and 28 interview participants) Specific Aim 2: Evaluate the impact of a half day mental health integrated emergency preparedness intervention in Pre-K-12 schools via shared leadership and peer support.
* Matched waitlist control comparison with 6 Pre-K-12 schools (N = 300) in a diverse school district. Data collected for all 6 schools at baseline, and two time points following the intervention.

The output of our project will be a curriculum manual and online toolkit for schools, including the resources necessary for schools to independently assess, implement and evaluate baseline levels of key outcomes and the impact of training content. Resources will be developed and disseminated to schools with the assistance of the Outreach Core, which has proven experience working with 15 school districts in our region. This project addresses NIOSH Emergency Preparedness and Response Cross-Sector Program Goal concerning safety climate (#1) and will specifically address two NIOSH NORA Healthy Work Design & Well-being objectives: #4: Reduce work organization-related chronic health conditions among workers and #6: Improve the safety, health, and well-being of workers through healthier work design and better organizational practices.

ELIGIBILITY:
Inclusion Criteria:

* Pre-K-12 schools, including school leadership, teacher, and staff

Exclusion Criteria:

* Schools other than Pre-K-12

Only adults are enrolled in this workforce-focused study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 519 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Psychological Preparedness (measuring change from pre to post intervention) | Immediately prior to intervention with follow-up approximately 2-4 weeks after the intervention is implemented
  This section has been adapted from existing sources. Examples of specific Psychological Preparedness Items are detailed below -
  * I am confident that I can perform the necessary actions in an emergency/high stress situation.
  * I am knowledgeable about the impact that emergencies/high stress situations can have on a person's ability to respond as they would like.
  All items are associated with a 5 point response scale from Strongly Disagree to Strongly Agree (higher scores = greater agreement). Individual items will be examined. A composite scale may be produced based on measures of internal consistency.
Emergency Preparedness Climate (measuring change from pre to post intervention) | Immediately prior to intervention with follow-up approximately 2-4 weeks after the intervention is implemented
  This section has been adapted from existing sources. Examples of specific Emergency Preparedness Climate Items are below -
  * My school provides a clear vision for emergency preparedness at work
  * My school tries to continually improve emergency preparedness
  All items are associated with a 5 point response scale from Strongly Disagree to Strongly Agree (higher scores = greater agreement). Individual items will be examined. A composite scale may be produced based on measures of internal consistency.
Shared leadership for Emergency Preparedness (measuring change from pre to post intervention) | Immediately prior to intervention with follow-up approximately 2-4 weeks after the intervention is implemented
  This section has been adapted from existing sources. Examples of specific Shared Leadership for Emergency Preparedness Items are below - School employees -
  * behave in a way that displays a commitment to emergency preparedness
  * provide a clear vision for emergency preparedness
  All items are associated with a 5 point response scale from Strongly Disagree to Strongly Agree (higher scores = greater agreement). Individual items will be examined. A composite scale may be produced based on measures of internal consistency.
Peer Support and Social Cohesion associated with Emergency Preparedness (measuring change from pre to post intervention) | Immediately prior to intervention with follow-up approximately 2-4 weeks after the intervention is implemented
  This section has been adapted from existing sources. Examples of specific Peer Support and Social Cohesion Items associated with Emergency Preparedness Items below - School employees -
  * help each other to prepare for emergencies in concrete ways
  * help each other to prepare for emergencies in emotionally supportive ways
  All items are associated with a 5 point response scale from Strongly Disagree to Strongly Agree (higher scores = greater agreement). Individual items will be examined. A composite scale may be produced based on measures of internal consistency.
Confidence in Emergency Preparedness (measuring change from pre to post intervention) | Immediately prior to intervention with follow-up approximately 2-4 weeks after the intervention is implemented
  All items related to 'confidence in district and school-level emergency preparedness' are below -
  * I am confident that my school district has prepared me to respond to a real emergency at my school.
  * I am confident that I can respond to a real emergency at my school.
  All items are associated with a response scale of not at all confident to very confident, 5 point scale (higher scores = greater confidence). Individual items will be examined. A composite scale may be produced based on measures of internal consistency.

SECONDARY OUTCOMES:
Stress/Work Stress (measuring change from pre to post intervention) | Immediately prior to intervention with follow-up approximately 2-4 weeks after the intervention is implemented
  All items related to 'perceived stress at work' are below - -Please check the number that describes how much stress/distress you have been experiencing in the past week, including today.
  Scale is 0-10 with 10 = greater stress/distress
  -Please share how much job-related stress you have been feeling in the past two weeks.
  Response scale is 5 point, from none to very much (higher scores = more stress). Individual items will be examined.
Depression (measuring change from pre to post intervention) | Immediately prior to intervention with follow-up approximately 2-4 weeks after the intervention is implemented
  All items related to 'depression' are below -
  * I have felt little interest or pleasure in doing things.
  * I have felt down, depressed, or hopeless.
    4-point scale: 1-not at all, 2-several, 3-more than half, 4-nearly every day (higher scores = greater symptoms). A composite scale may be produced based on measures of internal consistency.
Anxiety (measuring change from pre to post intervention) | Immediately prior to intervention with follow-up approximately 2-4 weeks after the intervention is implemented
  All items related to 'anxiety' are below -
  * I have felt nervous, anxious or on edge.
  * I have not been able to stop or control worrying.
  * I have been worrying too much about different things.
  * I have had trouble relaxing.
  * I have been so restless that it is hard to sit still.
  * I have become easily annoyed or irritable.
  * I have been feeling anxious about the potential for an emergency to happen at my job.
  * I have felt afraid, as if something awful might happen.
    4-point scale: 1-not at all, 2-several, 3-more than half, 4-nearly every day (higher scores = greater symptoms). Individual items will be examined. A composite scale may be produced based on measures of internal consistency.
Post-traumatic stress disorder (measuring change from pre to post intervention) | Immediately prior to intervention with follow-up approximately 2-4 weeks after the intervention is implemented
  All items related to 'PTSD' are below -
  * I have been feeling jumpy or easily startled
  * I have been having repeated, disturbing and unwanted memories of a stressful or traumatic event.
  * I have been avoiding external reminders of a stressful or traumatic event (for example, people, places, activities, conversations, activities, objects or situations).
  * I have been having strong negative beliefs about myself, other people or the world.
    4-point scale: 1-not at all, 2-several, 3-more than half, 4-nearly every day (higher scores = greater symptoms). Individual items will be examined. A composite scale may be produced based on measures of internal consistency.
Mental well-being (measuring change from pre to post intervention) | Immediately prior to intervention with follow-up approximately 2-4 weeks after the intervention is implemented
  Single item measure - How would you rate your overall mental health and wellbeing? Excellent, Very Good, Good, Fair, Poor, with higher scores indicating worse mental health
Burnout (measuring change from pre to post intervention) | Immediately prior to intervention with follow-up approximately 2-4 weeks after the intervention is implemented
  All items related to 'burnout' are below, adapted from existing measures. Considering this definition (definition provided), please share how much burnout you are feeling related to your job in the past two weeks.
  I have been thinking about quitting my job. I've been feeling optimistic about the future related to my job. I've been dealing with problems well at my job. I've been thinking clearly at my job. I've been feeling good about myself at my job.
  All items are associated with a 5 point response scale from Strongly Disagree to Strongly Agree (higher scores = greater agreement). Individual items will be examined. A composite scale may be produced based on measures of internal consistency.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Welton-Mitchell, PhD, Principal Investigator — Colorado School of Public Health
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
All participant survey data collected by the researchers will be made available in a timely manner upon written request.
Supporting Information: Study Protocol
Time Frame: The data will be available upon study completion in August 2023 and will be stored in the longer term for three years after the study concludes, per federal regulations.
Access Criteria: Files with de-identified data will be transferred via electronic format using a secure electronic file transfer along with a statement of data use standards. Documentation of data use standards will be included. To protect our participants we will make the data and its associated documentation available to users only under a data-sharing agreement that provides for:
  (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.